CLINICAL TRIAL: NCT02129803
Title: Evaluating High Flow Humidification Therapy in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20002205
Record Dates: First submitted 2014-04-10; First posted 2014-05-02 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, high flow 20 liters per minute (LPM) humidification therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Therapy (Experimental): High-Flow, 20 LPM (via Optiflow cannula) Heated (34C) Humidified Air
  Interventions: Device: High-Flow, 20 LPM (via Optiflow cannula)
- Control Therapy (Low Flow) (Placebo Comparator): Low FLow, 5 LPM (via Optiflow cannula) Room Temperature (23-26C) Ambient Air
  Interventions: Device: Low FLow, 5 LPM (via Optiflow cannula)

INTERVENTIONS:
Device: High-Flow, 20 LPM (via Optiflow cannula) — Nasal high flow humidification (20LPM) therapy will be administered using Optiflow with Airvo 2.
  Arms: Experimental Therapy
Device: Low FLow, 5 LPM (via Optiflow cannula) — standard humidified wall medical air.
  Arms: Control Therapy (Low Flow)

SUMMARY:
This study is a single center, randomized pilot study to evaluate the clinical effectiveness of nasal high flow 20LPM humidification therapy in subjects with Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Hospital admission for acute pulmonary exacerbation of CF (using Fuchs criteria 4/10)
* 10 years of age and older
* Subject is able to comply with the procedures scheduled in the protocol
* Signed informed consent form

Exclusion Criteria:

* Receipt of any aerosolized experimental or investigational drugs within 1 month of enrollment
* Subject had ear, nose, and throat (ENT) surgery, nasal bleeding, or nasal polyps within 6 months prior to study
* Subject is unlikely to comply with the procedures scheduled in the protocol
* Inability to give informed consent
* Subject requires supplemental oxygen
* History of obstructive sleep apnea
* History of pressure headaches requiring therapy within one month of enrollment
* Any other medical or psychological condition in which the study doctor(s) believe(s) would inhibit the individual from being an appropriate study subject.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Therapy | Control Therapy (Low Flow)
Started | 12 | 12
Completed | 6 | 9
Not Completed | 6 | 3
Not completed — Protocol Violation | 4 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Difficulty sleeping | 1 | 0
Not completed — Morning headache | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Therapy | Control Therapy (Low Flow) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (5.4) | 21.7 (6.7) | 20.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R)
Description: The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a validated health-related quality of life measure for CF that meets US Food and Drug Administration psychometric requirements for patient reported outcomes. It contains both generic and CF-specific scales and has demonstrated responsiveness in previous clinical studies. Scores range from 0 to 100 with higher scores indicating better health.
Time Frame: Day 0 to Day 6 or upon discharge from the hospital, whichever comes first
Population: Results could not be reported for 4 participants due to missing baseline data in one case, missing followup data in one case, and no CFQ-R data in two cases.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Experimental Therapy | Control Therapy (Low Flow)
Number analyzed (Participants) | 3 | 8
change in score on a scale
  Physical functioning subscale | 0.056 (0.105) | 0.052 (0.152)
  Vitality subscale | 0.192 (0.139) | 0.194 (0.115)
  Emotional state subscale | -0.089 (0.139) | 0.033 (0.087)
  Social limitations subscale | -0.056 (0.096) | -0.028 (0.154)
  Role limitations subscale | -0.056 (0.192) | 0.010 (0.175)
  Body image subscale | 0.037 (0.170) | 0.125 (0.192)
  Eating disturbances subscale | 0.037 (0.280) | 0.097 (0.162)
  Treatment constraints subscale | -0.037 (0.170) | -0.097 (0.093)
  Respiratory symptoms subscale | 0.019 (0.170) | -0.125 (0.856)
  Digestive symptoms subscale | 0.111 (0.192) | 0.028 (0.098)
  Weight subscale | -0.222 (0.192) | 0.083 (0.236)
  Health status subscale | -0.083 (0.399) | 0.000 (0.103)

2. Secondary Outcome: Sputum Collection
Description: Sputum is collected during pulmonary function test (PFT) to later measure the biophysical properties of cystic fibrosis sputum.
Time Frame: 10 minutes
Population: We were unable to collect sputum samples from the participants
Arm/Group | Experimental Therapy | Control Therapy (Low Flow)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Length of hospital stay - up to 3 months
Arm/Group | Experimental Therapy | Control Therapy (Low Flow)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 2/6 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Therapy (N=6) | Control Therapy (Low Flow) (N=9)
Nasal discomfort (Product Issues) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02129803/Prot_SAP_000.pdf